CLINICAL TRIAL: NCT00618735
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of BIIB021 Administered Once or Twice Daily to Subjects With Advanced Solid Tumors
Brief Title: Once or Twice Daily Administration of BIIB021 to Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120ST103
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — 6-chloro-9-(4-methoxy-3,5-dimethylpyridin-2-ylmethyl)-9H-purin-2-ylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subjects in Schedule A will take BIIB021 in the morning at approximately 0800 with at least 6 ounces of water following an overnight fast (Beginning at midnight).
  Interventions: Drug: BIIB021
- 2 (Experimental): Subjects in Schedule B will take BIIB021 in the morning at approximately 0800 with at least 6 ounces of water following an overnight fast (beginning at midnight). The second dose will be taken, following at least a 2-hour fast, 12 hours (+/- 2 hours) after the first dose, except on Day 1 of Cycle 1 and Day 1 of Cycle 2.
  Interventions: Drug: BIIB021

INTERVENTIONS:
Drug: BIIB021 — Dosage, frequency (once daily), and duration as specified in protocol. This dosing arm is currently on hold.
  Other Names: CNF2024
  Arms: 1
Drug: BIIB021 — Twice daily dosing
  Other Names: CNF2024
  Arms: 2

SUMMARY:
The purpose of the study is to see if daily and twice daily administration of BIIB021 is tolerated in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Heat shock protein 90 (HSP90) inhibitors are anticipated to have clinical activity in solid tumors because Hsp90 is required for the folding, activation, and assembly of many proteins involved in cancer cell survival, proliferation, and metastasis. The maximum tolerated dose (MTX) for BIIB021 administered twice weekly in a phase I study in subjects with advanced solid tumors have been defined at 600mg. It is now reasonable from a safety perspective and desirable from a pharmacokinetic perspective to evaluate more frequent dosing intervals in solid tumors with the goal of providing more sustained and completed inhibition of Hsp90.

ELIGIBILITY:
Inclusion Criteria:

Subjects with histologically or cytologically confirmed solid tumor who have failed or refused standard therapies or for which no approved therapy is available.

Age greater than or equal to 18 years at the time of informed consent. ECOG performance status of less than or equal to 2. Lab values consistent with adequate renal, hepatic, and bone marrow functions.

Exclusion Criteria:

Prior antitumor therapies, including prior experimental agents or approved antitumor small molecules and biologics within 28 days and all associated toxicities resolved to eligibility levels.

Subjects with known brain metastases. Concurrent severe or uncontrolled medical disease. Must utilize effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of BIIB021 | As specified in protocol

SECONDARY OUTCOMES:
PK and PD of BIIB021 | As specified in protocol
Antitumor activity | As specified in protocol

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Encinitas, California
  - Research Site, Santa Monica, California
  - Research Site, San Antonio, Texas

REFERENCES:
- [Background] Saif MW, Takimoto C, Mita M, Banerji U, Lamanna N, Castro J, O'Brien S, Stogard C, Von Hoff D. A phase 1, dose-escalation, pharmacokinetic and pharmacodynamic study of BIIB021 administered orally in patients with advanced solid tumors. Clin Cancer Res. 2014 Jan 15;20(2):445-55. doi: 10.1158/1078-0432.CCR-13-1257. Epub 2013 Oct 4. PMID 24097863